CLINICAL TRIAL: NCT03934047
Title: Visual Field Infiltration of Tranexamic Acid Reduced the Blood Loss in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-126
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: Visual Field Infiltration of Tranexamic Acid during the operation of total knee replacement.
  Interventions: Drug: Tranexamic Acid 100 MG/ML
- Group B (No Intervention): Group B: No Visual Field Infiltration of Tranexamic Acid during the operation of total knee replacement.

INTERVENTIONS:
Drug: Tranexamic Acid 100 MG/ML — Visual Field Infiltration of Tranexamic Acid during the operation of total knee replacement.
  Arms: Group A

SUMMARY:
Background and study aims Osteoarthritis (OA) is the most common type of arthritis, which most often affects the knee. It occurs when the protective cartilage on the end of bones wears away. The bones then rub against one another, which can cause stiffness, pain and a reduction in a person's range of movement. A knee joint replacement is a common procedure where the weight bearing surfaces of the knee joint are replaced with metal and plastic components to relieve the pain and disability brought on by OA. Tranexamic Acid（TXA） is a traditional method to reduce blood loss, pain score and complications. It is not known however, what is the best method of TXA for the patients with TKA. The aim of this study is to find out whetherVisual Field Infiltration of Tranexamic Acid Reduced the Blood Loss in patients who have had knee replacement surgery.

DETAILED DESCRIPTION:
Who can participate? Adults who have OA and need a total knee replacement. What does the study involve? Participants are randomly allocated to one of three groups. For the interventions field, could you please provide a brief methodology for each of your treatment arms, and the total duration of treatment and follow-up? Group A: Visual Field Infiltration of Tranexamic Acid during the operation of total knee replacement. Group B: No Visual Field Infiltration of Tranexamic Acid during the operation of total knee replacement.

The blood loss, VAS pain scores, length of their hospital stay, swelling and bleeding, and range of motion of the affected knee are assessed in the days following surgery.

What are the possible benefits and risks of participating? Participants who are allocated to receive treatment with Visual Field Infiltration of Tranexamic Acid may benefit from a reduction in blood loss, pain, swelling and blood loss after surgery, shortening their hospital stay.

There is a small risk of discomfort, frostbite or deep vein thrombosis (a blood clot in a major vein in the leg) when using Visual Field Infiltration of Tranexamic Acid.

ELIGIBILITY:
Inclusion Criteria:

Adults who have OA and need a total knee replacement.

Exclusion Criteria:

1. Patients had abnormal blood coagulation.
2. Patients were diagnosed as rheumatoid arthritis, traumatic osteoarthritis, ankylosing, spondylitis, hemophilic arthritis, peripheral vascular disease.
3. Cold urticaria.
4. Preoperative anticoagulation, patients had preoperative deep vein thrombosis (DVT).
5. Preoperative history of anemia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-26 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 1 week after operation
  Blood loss calculated by hemoglobin level

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided